CLINICAL TRIAL: NCT05659771
Title: Opportunities For Food Reformulation: Food Texture and Energy Density Effects on Eating Behaviour and Satiation
Brief Title: Opportunities for Food Reformulation
Acronym: OffR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: 4TU pride and prejudice project (Unknown)
Responsible Party: Principal Investigator, Marlou Lasschuijt, Assistant Professor, Wageningen University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: offR WUR
Record Dates: First submitted 2022-05-02; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Food; Energy Intake

STUDY DESIGN:
Intervention Model Description: The 5 conditions of this study are:
  1. low energy density, hard texture (slow eating rate)
  2. low energy density, soft texture (fast eating rate)
  3. High energy density, hard texture (slow eating rate)
  4. High energy density, soft texture (fast eating rate)
  5. Average energy density and medium hard texture (control)
Who Masked: Participant
Masking Description: cover story - different aim
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- low energy density, hard texture (Experimental): Sandwich with a hard texture (slow eating rate) and relatively low energy density (kcal/g)
  Interventions: Behavioral: Food properties manipulation to alter eating behavior and food and energy intake
- low energy density, soft texture (Experimental): Sandwich with a soft texture (fast eating rate) and relatively low energy density (kcal/g)
  Interventions: Behavioral: Food properties manipulation to alter eating behavior and food and energy intake
- High energy density, hard texture (Experimental): Sandwich with a hard texture (slow eating rate) and relatively high energy density (kcal/g)
  Interventions: Behavioral: Food properties manipulation to alter eating behavior and food and energy intake
- High energy density, soft texture (Experimental): Sandwich with a soft texture (fast eating rate) and relatively high energy density (kcal/g)
  Interventions: Behavioral: Food properties manipulation to alter eating behavior and food and energy intake
- Average energy density and medium hard texture (control) (Active Comparator): Sandwich with a medium texture (medium eating rate) and medium energy density (kcal/g)
  Interventions: Behavioral: Food properties manipulation to alter eating behavior and food and energy intake

INTERVENTIONS:
Behavioral: Food properties manipulation to alter eating behavior and food and energy intake — Food properties of commercially available food products

SUMMARY:
The objective of this study is to determine the independent and additive effects of food texture and energy density on food and energy intake compared to a control condition.

DETAILED DESCRIPTION:
Study design: The study has a 2x2 randomized crossover design. All participants receive 5 treatments and are their own control.

Study population: Healthy adults (n=75) between 18-55 years old with a BMI between 18.5-30 kg/m2.

Intervention: Participants will join 5 test days during which they receive, 5 test meals (lunch). The 5 test meals of this study are: 1.) low energy density, hard texture (slow eating rate) 2.) low energy density, soft texture (fast eating rate) 3.) High energy density, hard texture (slow eating rate) 4.) High energy density, soft texture (fast eating rate) 5.) Average energy density and medium hard texture (control). During eating and before and after eating the weight of the plate will be measured to determine intake. Additionally, participants will be recorded on video to determine eating behaviour (number of bites, chews and oral processing duration). The order in which participants will receive the diets will be randomized. The evening before and during each test day participants will keep a food and exercise diary.

Main study parameters/endpoints: The main study outcomes are food and energy intake of each lunch meal. Secondary outcomes are, eating behaviour characteristics measured by video (eating rate (g/min and bites/min), number of chews (chews/bite and chews/gram), bite size (gram/bite), oral processing duration (seconds), appetite (hunger, fullness, desire to eat, desire to eat sweet, desire to eat savoury, prospective consumption) and sensory characteristics (liking (taste + smell), desire to eat the meal, expected satiation, sweet, savoury, smoothness, chewiness, thickness) of the meals. Additional outcomes are individual differences in microstructure of eating, appetite responsiveness, eating Behavior phenotype, interoceptive sensitivity and anthropometry measures. During the trial new technology to capture food intake and eating behavior will be validated which is also an outcome of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-55 years old at the day of inclusion
* Able to understand and speak English fluently or without difficulty (self-report)
* BMI 18.5-30 kg/m2 - measured by the researchers at the end of information meeting
* Good general health and appetite ( self-report)
* Commonly (5 out of 7 week days) eating three meals a day every day around approximately the same times(Self-report).

Exclusion Criteria:

* Difficulties with swallowing, chewing and or eating in general
* Suffering from an endocrine or eating disorder, gastrointestinal illness or illness of the thyroid gland, respiratory disease or diabetes.
* Having taste or smell disorders (self-report)
* Braces (not including a dental wire) or oral piercing
* Smoking
* Consuming on average more than 21 glasses of alcohol per week (21)
* Not willing to stop using drugs during the study period (from inclusion till last test session)
* Use of medication that may influence study outcomes (self-report)
* Allergies or intolerance to any ingredient of the test meals or snacks
* Not willing to eat the test food because of eating habits, believes or religion.
* Following a vegetarian or vegan diet
* Lactose intolerant
* Men having facial hair such as a beard as facial movements cannot be analysed.
* Followed an energy restricted diet during the last 2 months
* Gained or lost 5 kg of body weight over the last half year
* High restrained eater according to the Dutch Eating Behaviour Questionnaire (men: score>2.89, women>3.39 )
* Signed up for participating in another research study
* Employee of Human Nutrition department of Wageningen university
* Thesis student or intern at the chair group of Sensory Science and Eating Behaviour Human Nutrition (WUR).
* Intensive exercising more than 8 hours per week
* Low score for liking the test foods on a nine point likert scale based on pictures of the food items.
* Unfamiliar with the test foods (self-report).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Energy intake | One meal, up to 30 minutes
  Intake in Kcal
Food intake | One meal, up to 30 minutes
  Intake in gram

SECONDARY OUTCOMES:
Eating rate | One meal, up to 30 minutes
  Eating rate gram/min
chews | One meal, up to 30 minutes
  number of chews per bite
bite size | One meal, up to 30 minutes
  gram/bite
Energy intake rate | One meal, up to 30 minutes
  kcal/min
bites | One meal, up to 30 minutes
  number of bites per meal
swallows | One meal, up to 30 minutes
  number of swallows per meal
oral exposure time | One meal, up to 30 minutes
  duration of food in mouth in seconds
Appetite | One meal, up to 30 minutes
  subjective ratings of appetite on a 100 mm line scale (visual analogue scale)
Individual differences in fat free mass (FFM) | 5 minutes
  % FFM of total body weight
individual eating rate | 1 minute
  eating rate (gram/min) of carrots of each participant (personal trait)
Individual appetite responsiveness | 10 minutes
  interoceptive sensitivity the ratio between the amount drank till first satiation signal and complete fullness, according to the waterload test
Sensory properties | 5 minutes
  rating on a 100mm line scale (visual analogue scale from 0 - not at all to 100 extremely) of the sensory properties of the sandwiches offered during the test sessions

OTHER OUTCOMES:
technology to measure intake automatically | One meal, up to 30 minutes
  automated weighing scales
technology to measure eating behavior | One meal, up to 30 minutes
  automated measures of eating behavior using video recordings

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen university, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lasschuijt MP, Heuven LA, Gonzalez-Estanol K, Siebelink E, Chen Y, Forde CG. The Effect of Energy Density and Eating Rate on Ad Libitum Energy Intake in Healthy Adults-A Randomized Controlled Study. J Nutr. 2025 Aug;155(8):2602-2610. doi: 10.1016/j.tjnut.2025.06.006. Epub 2025 Jun 12. PMID 40516651